CLINICAL TRIAL: NCT06717659
Title: Probiotics in the Management of Pulmonary Rehabilitation for COPD: a Randomized Controlled Trial
Brief Title: Probiotics in Pulmonaty Rehabilitation for COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Assistant Professor, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FJUH113385
Record Dates: First submitted 2024-11-24; First posted 2024-12-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Probiotic Intervention; Body Composition Measurement
Keywords: body composition; inflammation markers; nutritional supplementation; probiotics; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiotic group (Experimental): receive probiotics alongside standard pulmonary rehabilitation therapy
  Interventions: Other: probiotic supplementation intervention
- pulmonary rehabilitation group (Active Comparator): undergo only the standard pulmonary rehabilitation program
  Interventions: Other: standard pulmonnary rehabilitation

INTERVENTIONS:
Other: probiotic supplementation intervention — probiotic supplementation will be administered, while participants continue undergoing routine pulmonary rehabilitation therapy
  Arms: probiotic group
Other: standard pulmonnary rehabilitation — undergo routine pulmonary rehabilitation without probiotics intervention
  Arms: pulmonary rehabilitation group

SUMMARY:
This study aims to investigate various aspects of patients with chronic respiratory diseases undergoing pulmonary rehabilitation supplemented with probiotics. The focus will be on clinical physiological responses, functional performance, respiratory status assessments, nutritional status evaluations, body composition analyses, and biochemical blood parameters, with a primary emphasis on the anti-inflammatory response.

DETAILED DESCRIPTION:
Background： Patients with chronic obstructive pulmonary disease (COPD) often suffer from malnutrition and weight loss, which negatively impact mortality rates. Research indicates that insufficient intake of fiber, vitamins, and folic acid is associated with airflow limitation in COPD. Malnutrition affects lung function and muscle strength, leading to difficulty in breathing and reduced exercise tolerance. Nutritional support interventions, such as probiotics, are valuable in improving the nutritional status, lung function, and pulmonary rehabilitation in COPD patients.

Study Design： This is a one-year, single-center, prospective randomized controlled trial.

Methods： This study is a randomized controlled trial targeting COPD patients undergoing pulmonary rehabilitation. The plan is to recruit 60 participants, randomly assigned to either the probiotic intervention group or the conventional pulmonary rehabilitation group. The study includes physiological parameters, functional tests, questionnaires, and blood biochemical analyses. Data will be analyzed using SPSS, with statistical significance set at p < 0.05.

Effect： The trial expects that COPD patients receiving probiotic supplementation will achieve significant muscle gain and fat loss, reduce inflammation, and exhibit changes in body composition and functional performance.

Key words： Chronic obstructive pulmonary disease; probiotics; nutritional supplementation; inflammation markers; body composition

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign a written informed consent form.
* Diagnosed with pre-COPD or COPD stage I-IV according to the 2023 GOLD guidelines.
* Undergoing pulmonary rehabilitation therapy for more than three months.

Exclusion Criteria:

* Under 18 years old.
* Diagnosed with neuromuscular diseases.
* Experienced respiratory disease exacerbation requiring emergency care or hospitalization in the past three months.
* Unable to cooperate with cardiopulmonary exercise testing.
* Has other diseases or behavioral restrictions preventing participation in exercise training for over one year.
* Assessed by a physician to have severe malnutrition or a significantly low BMI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
interleukin-6 | six weeks
  inflammation evaluation

SECONDARY OUTCOMES:
indirect calorimetry | six weeks
  nutrition status
body composition analysis | six weeks
  nutrition status
heart rate | six weeks
  physiological parameters
saturation | six weeks
  physiological parameters
systolic and diastolic pressure | six weeks
  physiological parameters
respiratory rate | six weeks
  physiological parameters
six minute walk test | six weeks
  functional performance
time up and go | six weeks
  functional performance
FEV1 | six weeks
  functional performance
FVC | six weeks
  functional performance
FEV1/FVC | six weeks
  functional performance
CRP | six weeks
  biochemical blood tests
TNF-α | six weeks
  biochemical blood tests
TMAO | six weeks
  biochemical blood tests
The MDA of oxidative stress | six weeks
  biochemical blood tests
modified medical research council | six weeks
  self-perception questionnaire, maximun 4 and minimum 0, lower means a better outcome
COPD assessment test | six weeks
  self-perception questionnaire, maximun 40 and minimum 0, lower means a better outcome
Borg dyspnea scale | six weeks
  self-perception questionnaire, maximun 10 and minimum 0, lower means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No